CLINICAL TRIAL: NCT04406662
Title: Routine Evaluation of People Living With Cancer - Body Composition, Physical Function, Systemic Inflammatory Response, Quality of Life and Symptoms
Brief Title: Routine Evaluation of People Living With Cancer
Acronym: REVOLUTION
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC19154
Record Dates: First submitted 2020-03-13; First posted 2020-05-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Cachexia; Cancer; Advanced Cancer; Quality of Life
Keywords: cancer; advanced cancer; incurable cancer; body composition; physical function; symptoms; cachexia; quality of life; systemic inflammatory response; palliative medicine
MeSH Terms: conditions — Cachexia; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples - samples sent for routine inflammatory markers, plasma retained for analysis of cytokine levels and stored in a biobank for use in future ethically approved studies including potential genetic DNA analysis.
  Archival tissue specimens (including fresh frozen and/or formalin fixed paraffin embedded biopsy/surgical specimens) that are no longer required by the local pathologist for diagnostic purposes, or are stored as part of ethically approved tissue collection/research studies, may be requested from patients in the course of establishing the biobank for further analysis in future studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People with incurable cancer often have complex individual needs, however there are several common themes encountered when considering this group.

As cancer progresses there are series of interactions between the tumour and the patient, producing both local and systemic effects. This altered state of illness can have multiple ill effects including weight loss, fatigue, increased symptom burden and reduction in physical function which all contribute to a reduced quality of life.

These areas are often studied in isolation, giving an incomplete picture. A detailed, holistic characterisation of this group of people does not exist.

A robust characterisation of people with incurable cancer will allow identification and prioritisation of future research and has the potential to inform new therapeutics and provide justification for treatments.

This study aims to collect information about symptoms and quality of life, weight loss and body composition, physical activity and the body's immune response to cancer.

Participants with incurable cancer will be recruited to the study from oncology and palliative medicine services in the UK. Participants will answer questionnaires about quality of life and symptoms, have bloods taken for inflammatory marker and cytokine analysis and have their body composition measured by a variety of methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incurable cancer (metastatic cancer (Clinical, histological, cytological or radiological evidence) or receiving anti-cancer therapy with palliative intent).
* Aged 18-years and over
* Written informed consent

Exclusion Criteria:

* Any concomitant medical or psychiatric problems which, in the opinion of the investigator, would increase the risk of complication for the participant and/or investigator.
* Participants will not be able to take part in bio-impedance analysis if they have a pacemaker or implantable cardiac defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with incurable cancer recruited from oncology and palliative care services in the UK
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2029-08-08 (Estimated); Study Completion 2029-08-08 (Estimated)

PRIMARY OUTCOMES:
Association between inflammatory cytokines and clinical parameters in incurable cancer | 2 years
  Correlation of serum levels of inflammatory cytokines with clinical parameters including skeletal muscle mass, symptom based scores and physical activity as measured by actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Barry JA Laird, MBCHB MD, Principal Investigator — St Columba's Hospice/ University of Edinburgh
Locations (1):
- St Columba's Hospice, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Paval DR, Patton R, McDonald J, Skipworth RJE, Gallagher IJ, Laird BJ; Caledonian Cachexia Collaborative. A systematic review examining the relationship between cytokines and cachexia in incurable cancer. J Cachexia Sarcopenia Muscle. 2022 Apr;13(2):824-838. doi: 10.1002/jcsm.12912. Epub 2022 Jan 25. PMID 35080147